CLINICAL TRIAL: NCT00676858
Title: Gas Embolism With Use of Argon Plasma Coagulation
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Adnan Majid, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2008P000124
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Embolism, Air
Keywords: Embolism; Argon
MeSH Terms: conditions — Embolism, Air; Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to use transesophageal echocardiography (TEE) to determine the incidence, severity, and clinical significance of gas bubbles during argon plasma coagulation (APC).

DETAILED DESCRIPTION:
Gas embolism is a rare but serious complication of APC. We will use TEE to monitor for gas bubbles during APC. APC will be terminated if gas bubbles are associated with ischemic heart rhythms, wall motion abnormalities, or if large gas bubbles are noted in the left ventricle.

ELIGIBILITY:
Inclusion Criteria:

* Adults (male and female) 18 years of age or older
* Clinical indication for bronchoscopy (hemoptysis, airway obstruction, tumor excision, granulation tissue that is impairing endobronchial stent performance)
* Ability of the patient or proxy to read, comprehend, and sign informed consent document.

Exclusion Criteria:

* Presence of esophageal disorders that may complicate transesophageal echocardiography (strictures, varices, fistula, prior esophageal surgery)
* Presence of coagulopathy or other bleeding diathesis
* Inability to tolerate brief periods of apnea
* Presence of pulmonary vascular disease
* Pregnant women will not be included in this study because the potential fetal hypoxemia is not an acceptable risk.
* No exclusions will be made based on gender or race.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred to tertiary care center
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07-05 (Actual); Study Completion 2011-07-05 (Actual)

PRIMARY OUTCOMES:
incidence of gas bubbles with use of APC | end of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Majid, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD was not shared